CLINICAL TRIAL: NCT00169975
Title: Efficacy of the CMI Magnetocardiograph in Diagnosing Acute Coronary Syndromes in Patients Presenting With High Risk Unstable Angina as Defined by ACC/AHA Guidelines
Brief Title: Efficacy of the CMI Magnetocardiograph in Diagnosing Acute Coronary Syndromes in Patients Presenting With High Risk Unstable Angina.
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: CardioMag Imaging (Industry)
Responsible Party: Peter Smars, MD, Mayo Clinic
Other Study IDs: 738-04
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Magnetocardiograph — MCG and ECG recordings sequentially at the four pre-defined bed positions and watches the real-time magnetocardiogram traces on the computer screen. At each position, nine sensors record MCG data, thus forming a 3 x 3 point grid square with point-to-point separation of 40 mm. The number of cardiac cycles recorded at each position should be adequate for signal averaging. Recording time per position is typically 90 seconds. At the end of 4 sequential recordings, raw, unfiltered MCG data are stored.

SUMMARY:
A magnetocardiograph (MCG) is a device capable of recording of magnetic fields arising from the electrical activity of the heart with traces similar to an electrocardiogram (ECG). This system was developed as a noninvasive, non-contact diagnostics of obstructive coronary artery disease (CAD), and especially of lack of oxygen in the heart as in a heart attack. The overall objective of this study is to demonstrate the efficacy of this MCG device for the detection and diagnosis of lack of oxygen of the heart in patients with chest pain.

DETAILED DESCRIPTION:
Coronary Artery Disease is the leading cause of death in the United States. The non invasive detection of Acute Coronary Syndromes (ACS's) remains a clinical challenge. Electrocardiogram (ECG) may only diagnose myocardial infarction in 50 % of the cases. Magnetocardiography is a new and noninvasive method capable of measuring and mapping the magnetic field that is generated during the cardiac cycle. The electric current is affected by ischemic damage, which in turn alters the magnetic field. The magnetic field is not affected by body tissues, unlike the surface current measurements in ECG.

Comparisons: The diagnostic accuracy of the CMI-Magnetocardiograph will be compared to that of the ECG in diagnosing High Risk Unstable Angina.

ELIGIBILITY:
Inclusion criteria:

* Patients classified as having High Risk Unstable Angina according to the ACCIAHA guidelines.
* Age ≥ 18 years.

Exclusion criteria:

* Hemodynamically unstable patients.
* Patients who just prior to or just after admission exhibit tachycardia with heart rates exceeding 150 bpm.
* Patients with third degree AV Block.
* Patients with pacemakers or internal cardiac defibrillators.
* Patients who cannot lie in a supine position for the MCG examination.
* Patients who refuse entry into the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: *ACC/AHA Guidelines for Unstable Angina: High Risk (≥1 of the following)
  History
  * Accelerating tempo of ischemic symptoms in the last 48 hrs Pain
  * Prolonged, ongoing (>20 min) rest pain (resistant to treatment) Clinical findings
  * Pulmonary edema
  * New / ↑ MR murmur
  * S3 or new/ ↑ rales
  * Hypotension, brady -/tachycardia - Age>75y ECG
  * Angina at rest with transient ST changes >0.05 mV
  * New (L)BBB
  * Sustained VT Cardiac Markers
  * Markedly elevated troponin
  Patients classified as having high-risk unstable angina at presentation in the ED will be approached for enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2004-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
1. Determine the discriminatory ability of the scores derived from the MCG evaluation to discriminate between patients with versus without a clinical diagnosis of ACS at discharge. | 1 year
2. Compare the discriminatory ability of scores derived from the MCG, the troponin level, and the ECG results, separately or in combination, to discriminate between patients with without a diagnosis of ACS at discharge. | 1 year

SECONDARY OUTCOMES:
1. Evaluate the sensitivity of the MCG to detect an ultimate diagnosis of ACS, MI, CHF, or death at 1 month, 6 months, and 1 year following discharge. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Smars, M.D. EM, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States